CLINICAL TRIAL: NCT02657057
Title: Effects of Transcutaneous and Percutaneous Posterior Tibial Nerve Stimulation on Idiopathic Overactive Bladder Syndrome: Randomized Clinical Trial
Brief Title: Effects of Transcutaneous and Percutaneous PTNS on Idiopathic OAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Médico Tecnológico SL (Other)
Collaborators: University Ramon Llull (Other)
Responsible Party: Principal Investigator, Inés Ramírez García, Physiotherapist, MSc, Instituto Médico Tecnológico SL
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IMT46681770
Record Dates: First submitted 2015-12-20; First posted 2016-01-15 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Overactive Bladder; Urge Incontinence; Overactive Detrusor
Keywords: neuromodulation; electrical estimulation; percutaneous; transcutaneous; OAB
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transcutaneous Tibial Nerve Stimulation (Experimental): TENS SNS therapy is performed as follows; patient is asked to sit with legs slightly bent and an adhesive electrode is attached transcutaneously 5cm cephalic to either the right or left medial malleolus (subject choice). A surface electrode is placed on the medial surface of the ipsilateral calcaneum and both electrodes are connected to a low voltage electronic stimulator. The current is then set to the highest level tolerable to the subject (0-20 mA) and subject undergoes therapy for 30 minutes and 12 weeks (once-a-week session). Data are completed at baseline, after half therapy and after 12 weeks therapy.
  Interventions: Device: TENS SNS
- Percutaneous Tibial Nerve Stimulation (Active Comparator): PTNS therapy is performed as follows; patient is asked to sit with legs slightly bent. The area where the needle will be placed is cleaned with an alcohol swab. A 34 gauge needle (equivalent to an acupuncture needle) is inserted percutaneously approximately 5 cm cephalad to the medial malleolus of the right or left ankle (subject choice) at a 60 degree angle. A surface electrode is placed on the medial surface of the ipsilateral calcaneous. The needle and electrode are connected to a low voltage electrical stimulator. The current is then set to the highest level tolerable to the subject (0-20 mA) and the subject undergoes therapy for 30 minutes and 12 weeks (once-a-week session). Data are completed at baseline, after half therapy and after 12 weeks therapy.
  Interventions: Device: PTNS

INTERVENTIONS:
Device: PTNS — The needle and electrode are connected to a low voltage (9 V) electrical stimulator (URO stim2). Stimulation current with a fixed frequency of 20 Hz and a pulse width of 200 msec is increased until flexion of the big toe or fanning of all toes becomes visible, or until the subject reports a tingling sensation across the heel or bottom of the foot.
  Other Names: Percutaneous Tibial Nerve Stimulation (URO stim2)
  Arms: Percutaneous Tibial Nerve Stimulation
Device: TENS SNS — Electrodes are connected to a low voltage (9 V) electrical stimulator (URO stim2). Stimulation current with a fixed frequency of 20 Hz and a pulse width of 200 msec is increased until flexion of the big toe or fanning of all toes becomes visible, or until the subject reports a tingling sensation across the heel or bottom of the foot.
  Other Names: Transcutaneous Tibial Nerve Stimulation (URO stim2)
  Arms: Transcutaneous Tibial Nerve Stimulation

SUMMARY:
The purpose of this study is to determine if Transcutaneous Tibial Nerve Stimulation (TENS) is as effective as Percutaneous Tibial Nerve Stimulation (PTNS) as therapeutic option for subjects with Idiopathic Overactive Bladder (OAB) who have failed conventional therapy.

DETAILED DESCRIPTION:
Both therapies have been proven to be effective, but very few times have been compared. PTNS and TENS SNS have been proven effective modifying bladder diary scores (change in the frequency of day and night urination, and urge incontinence), and improving subject's quality of life. Only PTNS has shown changes in urodynamic data while undergoing therapy.

The investigators hypothesize that short-term effectiveness and benefit reported, is not lower in the TENS group, if we compare both therapies in a randomized control trial.

Secondary goals are to evaluate changes in bladder diary scores (frequency of urination, nocturia, number of urgency and leakage episodes ), participants quality of life improvement scores and treatment benefit score at TBS scale, while undergoing these therapies.

ELIGIBILITY:
Inclusion Criteria:

* Female and male
* Age >18 years
* Complaint urge urinary incontinence (3 or more episodes per week) OR overactive bladder (8 or more voids per day, and/or 2 or more voids per night)
* Urodynamic data of overactive detrusor
* Failed trial of conservative therapy (bladder training, fluid modification, diet modification, caffeine restriction, pelvic floor training)
* Failed trial of anticholinergic either due to inability to take the medication, adverse reaction to medication, or no improvement on medication
* Willing to complete study questionnaires and informed consent study

Exclusion Criteria:

* Presence of bladder obstruction (prostate or prolapse)
* Neurogenic bladder overactivity
* Previous pelvic organ prolapse surgery
* Unwilling and mentally incompetent to participate in study
* Pregnancy or planning to become pregnant during the study
* Presence of urinary fistula
* Recurrent or current urinary tract infection (5 or more infections in the last 12 months)
* Bladder stones
* Bladder cancer or suspected bladder cancer
* Hematuria
* Central or peripheral neurologic disorders such as Multiple Sclerosis, Parkinson's disease, spina bifida, or other spinal cord lesion
* Metal implants such as pacemaker, implantable defibrillator, or metal implants where PTNS or TENS device needs to be placed (sacrum or ankle/leg).
* Uncontrolled diabetes and diabetes with peripheral nerve involvement
* Anticoagulants treatment
* Current use of anticholinergics or use within the last 4 weeks
* Current use of botox bladder injections or bladder botox injection within the last year
* Current use of interstim therapy or currently implanted interstim device or leads
* Urinary retention or gastric retention
* Painful Bladder Syndrome/Interstitial Cystitis
* Previous PTNS treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2015-11; Primary Completion 2017-02 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Reduction from Baseline in Urinary Frequency Scores on 3-day voiding diaries at 12 weeks | 12 weeks
  A reduction in urinary frequency was regarded clinically significant when a normal voiding pattern of less than 8 voids per 24 hours could be obtained

SECONDARY OUTCOMES:
Reduction from Baseline in the number of leakage episodes diaries at 6 weeks and at 12 weeks | 6 and 12 weeks
  A reduction in the number of leakage episodes of at least 30% on 3-day voiding was regarded significant
Change from Baseline in Mean, Moderate to Severe Urgency episodes on 3-day voiding diaries at 6 and at 12 weeks | 6 and 12 weeks
  A reduction in number of urgency episodes at 6 weeks and 12 weeks
Reduction from Baseline in Mean Nocturia Episodes on 3-day voiding diaries at 6 and at 12 weeks | 6 and 12 weeks
  A reduction of at least 25% was regarded significant
Improved quality of life function via the Incontinence Quality of Life Scale (I-QOL) | 6 and 12 weeks
  An improvement of at least 10 points was regarded significant
Improved Bladder Symptom Severity Score via Overactive Bladder Questionnaire (OAB-q) at 6 and at 12 weeks | 6 and 12 weeks
  An improvement of at least 10 points was regarded significant
Degree of Satisfaction Score on the Treatment Benefit Scale (TBS) at 6 and at 12 weeks | 6 and 12 weeks
  A score of 1 or 2 was regarded significant

OTHER OUTCOMES:
Number of participants that request for continuous chronic treatment to keep the obtained response after receiving 12 PTNS/TENS sessions for OAB complaints | 12 weeks
  A number of at least 50% was regarded significant
Number of complaints OR adverse effects registered during treatments | From Baseline to week 12
  complaints and side effects were registered

CONTACTS AND LOCATIONS:
Overall Officials: Inés Ramírez, MSc, Principal Investigator — Instituto Médico Tecnológico
Locations (1):
- Inés Ramírez, Barcelona, Spain